CLINICAL TRIAL: NCT05834842
Title: An Internet-based Self-help Intervention for the Reduction of Consumption of Ultra-processed Products and Increase of Physical Activity in Mexican University Population: Study Protocol for a Randomized Controlled Trial
Brief Title: Online Intervention for Reduction of Ultra-processed Products and Increase of Physical Activity in University Students
Acronym: UNISALUD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Collaborators: Universidad de Colima (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNISALUD
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Physical Inactivity; Ultra Processed Food; Stress; Anxiety; Depression
MeSH Terms: conditions — Sedentary Behavior; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The study has two arms, one is the experimental group that receives the treatment and the other is the comparison group that will receive treatment after the 9 sessions of the experimental group finished. The patients in both groups will be evaluated pre and post/treatment. The participants are assigned randomly to the intervention or comparison group.
Who Masked: Participant
Masking Description: The patients are not aware that there is an experimental group and a control group, the participants are not related and do not know each other. The conditions of the study are only known by the researcher, the therapists, and the Research Ethics Committee of the Universidad de Guadalajara.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: Online Intervention Unisalud (Experimental): Participants in this group will receive 9 sessions of a multi-component intervention focused on the reduction of the consumption of ultra processed foods, symptoms of anxiety, depression and stress and the increase of physical activity.
  Interventions: Behavioral: Unisalud
- No Intervention: Waiting List group (No Intervention): The participants in this group will not receive the treatment, just waiting list. They will be measured one time and then a second time 3 months after. Calculating when 3 months corresponding to 9 sessions will receive the intervention.

INTERVENTIONS:
Behavioral: Unisalud — The "UNISALUD" intervention will be made up of 42 videos, made using the visual collage technique, where illustration, video fragments and visual interactions are mixed and in some there will be a presenter to achieve captivating visual material. to the participant. Likewise, it will be accompanied by digital infographics that will help reinforce the information proposed by the intervention.
  Arms: Behavioral: Online Intervention Unisalud

SUMMARY:
This study evaluates the effectiveness of an online Multi-component psychological intervention, that is focused on reducing the consumption of ultra processed foods and increase the frequency of performing Physical Activity. At the same time to observe the effect on symptoms of anxiety, depression and stress.

DETAILED DESCRIPTION:
Ultra Processed Products are edible products made primarily or entirely from substances derived from food. Its manufacture is based on industrial processes such as hydrogenation, extrusion and molding, pre-processed for frying, and that cannot be done at home. A sedentary lifestyle or physical inactivity is associated with loss of muscle mass and weight gain. In contrast, physical activity acts as a protector against non-communicable diseases such as type 2 diabetes, cardiovascular diseases and some types of cancer. AF levels are determined through Units of Measurement of the Metabolic Rate. Also the consumption of Ultra Processed Products and sedentary behaviors have been associated with affectations on people's health; An example of this is the association that exists between them and has been associated with an increased risk of suffering from depression, anxiety, and stress.

Internet-based interventions had a large effect on cognitive dietary outcomes, a moderate effect on dietary intake and weight, and a small effect on physical activity outcomes. In concrete, self-applied interventions can be an option to arrive at a great number of participants. In such intervention the user receives the treatment solely through a web platform or an App. Such interventions are usually composed of videos, text and audios. Different reviews regarding self-administered treatments via the internet and computer-based treatments have been found them to be effective to achieve their goals.

The intervention will follow the principles of User Experience, with this ensuring that the design characteristics of the tool will meet the desired requirements to be perceived as easy to use, attractive and useful.

This study will be conducted through a randomized controlled clinical superiority trial with two independent groups. It will include intra subjects at five evaluation moments: 1) pretest, 2) middle of the intervention, 3) post-test, 4) follow up at three months and 5) follow up at 6 months.

Participants will be randomly assigned to one of two groups: experimental group, "UNISALUD", composed of 9 sessions and interactive elements such as videos, audios and infographics; control group, will be the waiting list group, the participants in this group will not receive the treatment immediately, it will be measured one time and then a second time 27 days later than the experimental group when it is calculated that the first group has carried out the 9 sessions.

The measures will be the following:

1. Frequency of Consumption of ultra-processed foods
2. International Physical Activity Questionnaire
3. Health Action Process Approach
4. Self-Efficacy Eating Consumption Scale
5. Self-Efficacy Exercise Questionnaire
6. Stress Perception
7. Generalized Anxiety Disorder Scale
8. The Center for Epidemiological Studies Depression Scale
9. System Usability Scale

ELIGIBILITY:
Inclusion Criteria:

* Have a device (cell phone, computer or tablet) with internet access.
* Have agreed to participate by giving tacit consent.
* Be enrolled in any degree from a university in Mexico

Exclusion Criteria:

* Be diagnosed with a psychiatric disorder.
* Being diagnosed with an eating disorder.
* Being under some nutritional food treatment.
* Have a physical disability or injury that prevents you from engaging in mild to moderate physical activity.
* Being under any pharmacological treatment for a medical condition.
* Leaving the instruments unfinished.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the scores of the Frequency of Consumption | 1 to 1.5 months, depending on the development of the patient and the completion of the 9 modules
  To evaluate and monitor the consumption of PUs, a Consumption Frequency with emphasis on processing will be used, which was adapted from the Nova screener for the consumption of ultra-processed foods and the Consumption Frequency of foods of adolescents and adults (12 years or older), used in the National Health and Nutrition Survey, 2019, which shows the foods commonly consumed in Mexico. This is a qualitative instrument that evaluates the consumption of PUs in three categories: a) drinks (12 items); b) products that replace or accompany meals (26 items); and c) unhealthy snacks (12 items). Intake is reported on a previous day (yes or no) and in frequency of consumption per month (never, once a month, once every 15 days, and 1 to 7 times a week or more than once a day). The cut-off points were delimited based on previous studies: a) High consumption: 5 or more products per day, b) Medium consumption: between 2 and 4 products per day and c) Low one or non products
Change in time of the Physical Activity | 1 to 1.5 months, depending on the development of the patient and the completion of the 9 modules
  The short version of International Physical Activity questionnarie consists of 7 items and provides information about the time the person spends doing moderate and vigorous intensity activities, walking, and sitting in the last seven days. The questionnaire classifies the level of activity carried out into three categories: low, moderate and high
Change in the Scale in Self- Efficacy Eating Consumption Scale (SEECS) | 1 to 1.5 months, depending on the development of the patient and the completion of the 9 modules
  Self-Efficacy Eating consumption Scale, consisted of 21 items with a response option ranging from 1 to 10, where 1 represents the absence of capacity and 10 represents being very capable of reducing the intake of caloric products or sweets and change the consumption of healthy foods. In addition, they were asked if they engaged in any type of physical activity. This scale shows reliability criteria of (α = 0.93).
Change in the Self-Efficacy for Exercise Questionnaire (SEEQ) | 1 to 1.5 months, depending on the development of the patient and the completion of the 9 modules
  The Self- Efficacy for Exercise Questionnaire assesses the degree of confidence that people perceive to be physically active. The full scale is composed of 5 items that assess negative affect, resistance to relapse, and giving oneself time to be physically active. It is Likert-type and its response options range from 1 (not at all confident) to 5 (extremely confident).
Change in the Sedentary behavior questionnarie (SBQ-s) | 1 to 1.5 months, depending on the development of the patient and the completion of the 9 modules
  The SBQ-s has 11 items that assess the time spent on sedentary behaviors (e.g., watching television, eating while sitting, resting while lying down, driving or traveling by car, bus, or subway). These activities are evaluated on both a typical weekday and a weekend day. The response options are: "none," "15 minutes or less," "30 minutes," "1 hour," "2 hours," "3 hours," "4 hours," "5 hours," and "more than 6 hours." The time dedicated to each activity is converted into hours.

SECONDARY OUTCOMES:
Change in the Perceived Stress Scale | 1 to 1.5 months, depending on the development of the patient and the completion of the 9 modules
  Culturally the Perceive Stress Scale it has been adapted in Mexico by González-Ramírez & Landero-Hernández (2007). It is a Likert-type of 14 items with response options to 0 (never) to 4 (very often) to evaluate the degree to which situations in one's life are appraised as stressful.
Change in the Generalized Anxiety Disorder Scale (GAD-7) | 1 to 1.5 months, depending on the development of the patient and the completion of the 9 modules
  It is Likert-type of seven ítems and its response options range from 0 (not at all) - 3 (nearly every day). A score between 0 and 3 points indicates no perceived anxiety, and a score between 15 and 21 is an indicator of severe perceived anxiety
Change in the Center for Epidemiological Studies Depression Scale (CES-D) | 1 to 1.5 months, depending on the development of the patient and the completion of the 9 modules
  It was designed based on the study of clinical and general populations, and is currently one of the most widely used to assess depressive symptomatology in clinical and research settings at international and national level. It consists of 35 questions and contains five possible answers ranging from "Scarcely" (0 to 1 day), "Somewhat" (1-2 days), "Occasionally" (3-4 days), "Most" (5-7 days) and "Almost daily" (10-14 days).

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Dominguez Rodriguez, PhD, Study Chair — ITLAS group; Itzel Refugio Alvarado-Ávalos, BD, Study Chair — University of Guadalajara; Fátima López-Alcaraz, PhD, Study Chair — Universidad de Colima; Estefania Gasca-Suarez, BD, Study Chair — University of Guadalajara; Adrian Antonio Cisneros-Hernández, PhD, Study Chair — University of Guadalajara; Alexandra Valadez, PhD, Study Chair — University of Guadalajara; Fabiola Macías-Espinoza, PhD, Study Chair — University of Guadalajara

IPD SHARING:
Plan to Share IPD: Yes
The information will be available in a private server or in a server of the journal(s) that we will publish the articles that will be the result of this study. The protocol of the study is currently in progress to be published, in this article will be included such study protocol, the informed consent is already shared in the register of clinical trials.
Supporting Information: ICF
Time Frame: This data will be available approximately in February 2024 and it will be permanently available. It will be shared in the databases of the journal where the article(s) will be published.
Access Criteria: Through the servers of the journal(s) where we will publish the articles.

REFERENCES:
- [Background] Bhutani S, Cooper JA. COVID-19-Related Home Confinement in Adults: Weight Gain Risks and Opportunities. Obesity (Silver Spring). 2020 Sep;28(9):1576-1577. doi: 10.1002/oby.22904. Epub 2020 Aug 6. No abstract available. PMID 32428295
- [Background] Belogianni K, Baldwin C. Types of Interventions Targeting Dietary, Physical Activity, and Weight-Related Outcomes among University Students: A Systematic Review of Systematic Reviews. Adv Nutr. 2019 Sep 1;10(5):848-863. doi: 10.1093/advances/nmz027. PMID 31181143
- [Background] Dominguez-Rodriguez A, De La Rosa-Gomez A. A Perspective on How User-Centered Design Could Improve the Impact of Self-Applied Psychological Interventions in Low- or Middle-Income Countries in Latin America. Front Digit Health. 2022 Jun 2;4:866155. doi: 10.3389/fdgth.2022.866155. eCollection 2022. PMID 35721795
- [Background] Marino M, Puppo F, Del Bo' C, Vinelli V, Riso P, Porrini M, Martini D. A Systematic Review of Worldwide Consumption of Ultra-Processed Foods: Findings and Criticisms. Nutrients. 2021 Aug 13;13(8):2778. doi: 10.3390/nu13082778. PMID 34444936
- [Background] López-Torres, L. P., & López-Alcaraz, F. (2022). Los productos ultra-procesados: Implicancias sobre su consumo, avances y retos en América Latina para la salud pública en adultos (Ultra-processed products: Implications for their consumption, advances and challenges in Latin America for public health in adults). Revista chilena de nutrición, 49(5), 637-643.
- [Background] Castro O, Bennie J, Vergeer I, Bosselut G, Biddle SJH. How Sedentary Are University Students? A Systematic Review and Meta-Analysis. Prev Sci. 2020 Apr;21(3):332-343. doi: 10.1007/s11121-020-01093-8. PMID 31975312
- [Result] Medina C, Barquera S, Janssen I. Validity and reliability of the International Physical Activity Questionnaire among adults in Mexico. Rev Panam Salud Publica. 2013 Jul;34(1):21-8. PMID 24006016
- [Result] Palacios, J., Ramírez, V., Anaya, M., Hernández, H. L., & Martínez, R. (2017). Evaluación psicométrica de una escala de autoeficacia de la conducta alimentaria (Psychometric evaluation of a self-efficacy scale of eating behavior). Revista chilena de nutrición, 44(1), 95-102.
- [Result] Marcus BH, Selby VC, Niaura RS, Rossi JS. Self-efficacy and the stages of exercise behavior change. Res Q Exerc Sport. 1992 Mar;63(1):60-6. doi: 10.1080/02701367.1992.10607557. PMID 1574662
- [Result] Ramirez MT, Hernandez RL. Factor structure of the Perceived Stress Scale (PSS) in a sample from Mexico. Span J Psychol. 2007 May;10(1):199-206. doi: 10.1017/s1138741600006466. PMID 17549893
- [Result] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Result] Gonzalez-Forteza C, Jimenez-Tapia JA, Ramos-Lira L, Wagner FA. [Application of the revised version of the Center of Epidemiological Studies Depression Scale in adolescent students from Mexico City]. Salud Publica Mex. 2008 Jul-Aug;50(4):292-9. doi: 10.1590/s0036-36342008000400007. Spanish. PMID 18670720
- [Derived] Gonzalez-Cantero JO, Lopez-Torres LP, Alvarado-Avalos IR, Lopez-Alcaraz F, Gasca-Suarez E, Cisneros-Hernandez AA, Valadez A, Macias-Espinoza F, Dominguez-Rodriguez A. An internet-based self-help intervention for the reduction of consumption of ultra-processed products and increase of physical activity in Mexican university population: study protocol for a randomized controlled trial. Front Nutr. 2024 Jul 29;11:1325528. doi: 10.3389/fnut.2024.1325528. eCollection 2024. PMID 39221160

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-04-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT05834842/Prot_ICF_000.pdf